CLINICAL TRIAL: NCT00888745
Title: A Phase I, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Pharmacokinetics of PRO283698 in Patients With Rheumatoid Arthritis
Brief Title: A Study of the Safety and Pharmacokinetics of PRO283698 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Disclosures Group, Genentech, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: []4623g
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Rheumatoid Arthritis
Keywords: RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — pateclizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: PRO283698
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Intravenous and subcutaneous ascending dose
  Arms: 2
Drug: PRO283698 — Intravenous and subcutaneous ascending dose
  Arms: 1

SUMMARY:
This is a Phase I multicenter study that will be conducted in the United States and Europe.

ELIGIBILITY:
Inclusion Criteria:

* RA diagnosed according to the American College of Rheumatology (ACR)

Exclusion Criteria:

* Female patients who are pregnant, plan to become pregnant during the study, or are breastfeeding
* Clinically significant abnormal ECG
* History of anaphylactic reactions
* Positive hepatitis C antibody or hepatitis B surface antigen
* Positive serology for human immunodeficiency virus (HIV) by quantitative polymerase chain reaction
* A history of an autoimmune disease other than RA (other than secondary Sjogren syndrome)
* Significant systemic involvement of RA, including vasculitis, pulmonary fibrosis, or Felty syndrome
* Malignancy, or prior malignancy, other than non-melanoma skin cancer, or cervical carcinoma in situ that has been resected
* Recent administration of a live, attenuated vaccine, or anticipation that such a live attenuated vaccine will be required during the study or within 60 days after the last dose
* Concomitant therapy with a biologic agent
* Recent exposure to any investigational agent
* Any current or recent signs or symptoms of infection requiring parenteral antibiotic administration
* Hospitalization for a clinically relevant event within the 4 weeks prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of PRO283698 assessed through the incidence of adverse events | Through study completion or early study discontinuation

SECONDARY OUTCOMES:
Pharmacokinetic parameters | Following study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: June Lee, M.D., Study Director — Genentech, Inc.
Locations (12):
- United States (9):
  - Investigational Site, Anniston, Alabama
  - Investigational Site, Orlando, Florida
  - Investigational Site, Ormond Beach, Florida
  - Investigational Site, Palm Harbor, Florida
  - Investigational Site, Idaho Falls, Idaho
  - Investigational Site, Indianapolis, Indiana
  - Investigational Site, Frederick, Maryland
  - Investigational Site, Oklahoma City, Oklahoma
  - Investigational Site, Duncansville, Pennsylvania
- Hungary (3):
  - Investigational Site, Budapest
  - Investigational Site, Debrecen
  - Investigational Site, Szeged

REFERENCES:
- [Derived] Emu B, Luca D, Offutt C, Grogan JL, Rojkovich B, Williams MB, Tang MT, Xiao J, Lee JH, Davis JC. Safety, pharmacokinetics, and biologic activity of pateclizumab, a novel monoclonal antibody targeting lymphotoxin alpha: results of a phase I randomized, placebo-controlled trial. Arthritis Res Ther. 2012 Jan 8;14(1):R6. doi: 10.1186/ar3554. PMID 22225620